CLINICAL TRIAL: NCT02918721
Title: A Randomised, Multi-center, Subject and Evaluator-blinded Study Comparing Pain and Safety Profile Associated With Correction of Moderate to Severe Nasolabial Folds Using Restylane With and Without Addition of 0.3% Lidocaine Hydrochloride
Brief Title: Pain and Safety of Restylane With and Without Lidocaine for Correction of Moderate and Severe Nasolabial Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 43CH1504
Record Dates: First submitted 2016-09-22; First posted 2016-09-29 (Estimated); Results first posted 2021-01-06 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Nasolabial Fold
Keywords: Hyaluronic Acid, Nasolabial Fold, Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restylane Lidocaine (Experimental): Restylane Lidocaine will be injected into one side nasolabial fold on Day 1
  Interventions: Device: Restylane Lidocaine
- Restylane (Active Comparator): Restylane will be injected into the opposite side nasolabial fold on Day 1
  Interventions: Device: Restylane

INTERVENTIONS:
Device: Restylane Lidocaine — Intradermal injection
  Arms: Restylane Lidocaine
Device: Restylane — Intradermal injection
  Arms: Restylane

SUMMARY:
The purpose of this study is to evaluate the pain and safety associated with injections of Restylane Lidocaine compared to Restylane using a visual analogue scale.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Men or women aged 18 years or older of Chinese origin
* Subjects willing to abstain from any other facial plastic surgical or cosmetic procedures below the level of the lower orbital rim for the duration of the study
* Intent to undergo correction of both nasolabial folds(NLF) with a wrinkle severity in Wrinkle Severity Rating Scale(WSRS) of either 3 on both sides or 4 on both sides

Exclusion Criteria:

* Previous use of any permanent (non-biodegradable) or semi-permanent facial tissue augmentation therapy or autologous fat below the level of the lower orbital rim
* Previous use of any hyaluronic acid based or collagen based biodegradable facial tissue augmentation therapy below the level of the lower orbital rim within 12 months before treatment
* Previous tissue revitalisation treatment with laser or light, mesotherapy radiofrequency, chemical peeling or dermabrasion in the midface within 6 months before treatment
* Scars or deformities, active skin disease, inflammation or related conditions near or in the area to be treated
* Other condition preventing the subject from entering the study in the Investigator's opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2017-04-27 (Actual); Study Completion 2017-05-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Q-Med AB, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 70 subjects enrolled and each subject has 2 NLFs, in total 70 NLFs were injected with Rstylane, opposite 70 NLFs was Restylane Lido.
Groups:
- All Study Participants: Restylane Lidocaine will be injected into one side of the nasolabial fold at day 1 Restylane Lidocaine: Intradermal injection Restylane will be injected into the opposite side of the nasolabial fold on day 1 Restylane: Intradermal injection
Period: Overall Study
Arm/Group | All Study Participants
Started | 70
Completed | 70
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Han Chinese | 70
Region of Enrollment [Number; unit: participants]
  China | 70

OUTCOME MEASURES:

1. Primary Outcome: Treatment Difference in Pain (Restylane Lidocaine Side - Restylane Side) as Measured by a Visual Analogue Scale(VAS)
Description: Subjects that reported at least 10 mm less VAS pain associated with injections of Restylane-Lido compared to Restylane at the time of injection.
  VAS=Visual Analogue Scale. The VAS is a subjective scale to measure pain intensity. The participant is instructed to put a vertical mark, approximating the pain experienced during the procedure, on a 100 mm (millimeter) horizontal line labelled "no pain" at the left end and "the worst pain you can imagine" at the right end. The distance in mm from the left end (no pain) to the participant's VAS mark is measured with a standard ruler.
Time Frame: Up to 60 minutes after Injection on Day of Treatment
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- All Study Participants: Restylane Lidocaine will be injected into one side nasolabial fold on Day 1
  Restylane Lidocaine: Intradermal injection
  Restylane will be injected into opp side nasolabial fold on Day 1
  Restylane: Intradermal injection
Arm/Group | All Study Participants
Number analyzed (Participants) | 70
percentage of subjects | 77.1 [65.6 to 86.3]

2. Secondary Outcome: Treatment Differences in Pain (Restylane Side - Restylane Lidocaine Side) as Measured by a Visual Analogue Scale (VAS)
Description: Subjects that reported at least 10 mm less VAS pain associated with injections of Restylane-Lido compared to Restylane at 15, 30, 45 and 60 minutes after injection. VAS=Visual Analogue Scale. The VAS is a subjective scale to measure pain intensity. The participant is instructed to put a vertical mark, approximating the pain experienced during the procedure, on a 100 mm (millimeter) horizontal line labelled "no pain" at the left end and "the worst pain you can imagine" at the rig
Time Frame: 15, 30, 45, and 60 minutes after injection
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | All Study Participants
Number analyzed (Participants) | 70
percentage of subjects
  after 15 minutes | 55.7 [43.3 to 67.6]
  after 30 minutes | 48.6 [36.4 to 60.8]
  after 45 minutes | 35.7 [24.6 to 48.1]
  after 60 minutes | 31.4 [20.9 to 43.6]

ADVERSE EVENTS:
Time Frame: Up to 2 weeks
Description: Each subject was asked about AEs at each clinical visit. The question asked was "Since your last clinical visit have you had any health problems?". Information on AEs could also be obtained from signs and symptoms detected during each examination or from a laboratory test, observations by the study personnel, subject diaries or spontaneous reports from the subjects.
Groups:
- All Study Participants: Restylane Lidocaine will be injected into one side nasolabial fold on Day 1
  Restylane Lidocaine: Intradermal injection
  Restylane will be injected into one side nasolabial fold on Day 1
  Restylane: Intradermal injection
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70
Other Adverse Events (participants affected / at risk) | 8/70
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=70)
Pyrexia (Gastrointestinal disorders) | 1 (1)
Food allergy (Immune system disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Immune system disorders) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) — This contusion occurred on other parts of body but not nose side.
Alanine aminotransferase increased (Investigations) | 1 (1)
Blood uric acid increased (Investigations) | 1 (1)
Transaminases abnormal (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-06-15): https://cdn.clinicaltrials.gov/large-docs/21/NCT02918721/Prot_002.pdf
  • Statistical Analysis Plan (2016-05-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT02918721/SAP_003.pdf